CLINICAL TRIAL: NCT07111156
Title: A Randomized, Double-Blind, Three-Arm, Prospective, Single-Center Clinical Study to Evaluate the Safety, Efficacy, and Tolerability of Pinorox® in Subjects With Facial Signs of Aging
Brief Title: A Clinical Study to Test the Safety and Effectiveness of Pinorox® for Improving Visible Signs of Facial Aging Such as Wrinkles, Fine Lines, and Dark Spots.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Ambe Phytoextracts Pvt. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NB250027-AP_1.0_08Jul25
Record Dates: First submitted 2025-07-17; First posted 2025-08-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-07

CONDITIONS: Fine Lines; Wrinkles; Facial Sign of Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical Cream containing 0.1% Pinorox® (Experimental): Mode of Usage: Apply a coin size (approximately 1g) amount of the test treatment to the face and gently massage it until fully absorbed.
  Frequency: Apply the treatment twice daily Route of administration: Topical Dosage Form: Semisolid (Cream) Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight.
  Interventions: Other: Topical Cream containing 1% Pinorox®; Other: Placebo (Base Cream)
- Topical Cream containing 1% Pinorox® (Experimental): Mode of Usage: Apply a coin size (approximately 1g) amount of the test treatment to the face and gently massage it until fully absorbed.
  Frequency: Apply the treatment twice daily Route of administration: Topical Dosage Form: Semisolid (Cream) Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight.
  Interventions: Other: Topical Cream containing 0.1% Pinorox®; Other: Placebo (Base Cream)
- Placebo (Base Cream) (Placebo Comparator): Mode of Usage: Apply a coin size (approximately 1g) amount of the test treatment to the face and gently massage it until fully absorbed.
  Frequency: Apply the treatment twice daily Route of administration: Topical Dosage Form: Semisolid (Cream) Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight.
  Interventions: Other: Topical Cream containing 0.1% Pinorox®; Other: Topical Cream containing 1% Pinorox®

INTERVENTIONS:
Other: Topical Cream containing 0.1% Pinorox® — Mode of Usage: Apply a coin size (approximately 1g) amount of the test treatment to the face and gently massage it until fully absorbed.
  Frequency: Apply the treatment twice daily Route of administration: Topical Dosage Form: Semisolid (Cream) Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight.
  Arms: Placebo (Base Cream); Topical Cream containing 1% Pinorox®
Other: Topical Cream containing 1% Pinorox® — Mode of Usage: Apply a coin sized (approximately 1 g) amount of the test treatment to the face and gently massage it until fully absorbed.
  Frequency: Apply the treatment twice daily Route of administration: Topical Dosage Form: Semisolid (Cream) Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight.
  Arms: Placebo (Base Cream); Topical Cream containing 0.1% Pinorox®
Other: Placebo (Base Cream) — Mode of Usage: Apply a coin sized (approximately 1 g) amount of the test treatment to the face and gently massage it until fully absorbed.
  Frequency: Apply the treatment twice daily Route of administration: Topical Dosage Form: Semisolid (Cream) Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight.
  Arms: Topical Cream containing 0.1% Pinorox®; Topical Cream containing 1% Pinorox®

SUMMARY:
A Randomized, Double-Blind, Three-Arm, Prospective, Single-Center Clinical Study to Evaluate the Safety, Efficacy, and Tolerability of Pinorox® in Subjects with Facial Signs of Aging

DETAILED DESCRIPTION:
This is a randomized, double-Blind, three-arm, prospective, single-centre clinical study to evaluate the safety, efficacy, and tolerability of pinorox® in subjects with facial signs of aging. A total of 81 subjects (27 subjects/treatment) will be enrolled in the study, comprising male and non-pregnant, non-lactating female participants aged 35 to 55 years (inclusive). Subjects must present with visible Crow's feet wrinkles, fine lines, and facial dark spots at baseline. Participants will be equally distributed across three treatment groups with 27 subjects per group.

The study is designed to complete with at least 75 evaluable subjects (25 per treatment group), accounting for potential dropouts or withdrawals during the study period.

The potential subjects will be screened as per the inclusion and exclusion criteria only after obtaining the written informed consent from the study participants. Subjects will be contacted telephonically by recruiting department prior the enrolment visit.

There will be total of 3 visits during the study. The duration of the study will be 60 Days (8 weeks) from the enrolment. Subjects will be instructed to visit the facility as per below visits.

Visit: 01 (Day 01, Week 00): Screening, ICD obtained, Enrolment, Baseline readings and post product usage readings.Visit 02 (Day 30, Week 04): Treatment Phase, Evaluations Visit 03 (Day 60, Week 08): Evaluations and Treatment Phase end | End of Study

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 35 to 55 years (both inclusive) at the time of consent. 2) Sex: Adult male and female having Crow's feet area wrinkles, fine lines, facial dark spots.

  3) Females of childbearing potential should have a self-reported negative urine pregnancy test at the time of screening visit.

  4) Subjects should not have used any cosmetic, nutraceutical or therapeutic products for skin ageing in last 3 months.

  5) Subjects are not allowed to participate in any other study until this study is complete.

  6) Subjects must be willing and able to follow the study directions and to return for all specified visits with the product.

  7) Subjects must agree to record each use of the test products in the subject's diary card on daily basis.

  8) Subjects must agree to record medication use during the study

Exclusion Criteria:

* 1) Subjects who are on steroids for last six months. 2) Subjects who have used any cosmetic, nutraceutical or therapeutic products for skin last three months.

  3) Subjects who are on product which contains kojic acid, glycolic acid, niacinamide, alpha arbutin, Vitamin C and other skin ageing product.

  4) Subjects with other dermatologic diseases whose presence or treatments could interfere with the assessment of study.

  5) Subjects that are pregnant and/or breastfeeding. 6) The subject has a known allergy or sensitivity to soaps, lotions, detergents, detanglers or fragrances.

  7) Subjects if do not agree to limit sun exposure to affected areas such as face during prolonged sun exposure.

  8) The subject has any other skin conditions i.e. cuts, scratches, ring worms, etc. which in the opinion of the Investigator, will interfere with the study results or will create undue risk for the subject.

  9) The subject has any of the conditions or factors that the Investigator believes may affect the response of the skin or the interpretation of the test results.

  10) The subject is currently taking or has taken any medication, which the Investigator believes may influence the interpretation of the data.

  11) Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-02-17 (Estimated); Study Completion 2026-02-17 (Estimated)

PRIMARY OUTCOMES:
Change in skin texture i.e. Crow's feet area wrinkles, fine lines, pores, roughness, dryness, smoothness | baseline on Day 01 (prior to the treatment usage) to post treatment assessments on Day 01 after 30 mins, Day 30 and Day 60
  evaluated through Visioscan VC 20 Plus, Crow's feet area wrinkles (score 0-3, score 0 indicate no wrinkles, score 3 indicate severe wrinkles), fine lines, pores, roughness, dryness, smoothness (measure in %)
Change in skin elasticity (R2) and firmness (RO) | from baseline on Day 01 (prior to the treatment usage) to post treatment assessments on Day 01 after 30 mins, Day 30 and Day 60
  evaluated through Cutometer Dual MPA 580 (R0 and R2) (change in %)
Change in skin pigmentation and dark spots | baseline on Day 01 (prior to the treatment usage) to post treatment assessments on Day 01 after 30 mins, Day 30 and Day 60
  evaluated through Mexameter MX 18 (change in %)
Change in skin colour parameters - L*, a*, b*, and ITA | baseline on Day 01 (prior to the treatment usage) to post treatment assessments on Day 01 after 30 mins, Day 30 and Day 60
  evaluated through Skin Colorimeter CL 400, L*, a*, b*, and ITA measure in change in %

SECONDARY OUTCOMES:
Change in skin dryness, redness, fine wrinkling/lines, coarse wrinkles, laxity, roughness and sallowness | from baseline on Day 01 (prior to the treatment usage) to post treatment assessments on Day 01 after 30 mins, Day 30 and Day 60
  evaluated through PGA scoring using Griffiths scale (minimum score 0- No appearance and maximum score 7-9- severe)
Change in skin wrinkles and fine lines | from baseline on Day 01 (prior to the treatment usage) to post treatment assessments on Day 01 after 30 mins, Day 30 and Day 60
  evaluated through Glogau skin age classification (Type I to Type IV based on wrinkles) Measure changes in %
Change in skin pigmentation | from baseline on Day 01 (prior to the treatment usage) to post treatment assessments on Day 01 after 30 minutes, Day 30 and Day 60
  evaluated through Melasma Area and Severity Index (MASI)(Changein %)
Change in skin hydration | from baseline on Day 01 (prior to the treatment usage) to post treatment assessments on Day 01 after 30 minutes, Day 30 and Day 60
  evaluated through Corneometer (change in %)
Change in skin glow | from baseline on Day 01 (prior to the treatment usage) to post treatment assessments on Day 01 after 30 minutes, Day 30 and Day 60
  evaluated through skin Glossymeter (Change in %)
Change in facial photographs | from baseline on Day 01 (prior to the treatment usage) to post treatment assessments on Day 30 (±2 Days) and Day 60 (±2 Days),
  through digital photography by Nikon Digital Camera D3300 or Similar
Change in product perception questionnaire | from baseline on Day 01 (prior to the treatment usage) to post treatment assessments on Day 30 and Day 60
  regarding change in dark spots, skin appearance, skin hydration, skin texture, reduced fine lines and wrinkles evaluated through 5-point Likert Scale (1-minimum score and 5-maximum score)

CONTACTS AND LOCATIONS:
Overall Officials: Nayan Patel, Principal Investigator — Study Principal Investigator
Locations (1):
- NovoBliss Research Private Limited, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No